CLINICAL TRIAL: NCT02807428
Title: A Phase 2 Randomized Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of a Single Intrathecal Preoperative Administration of AYX1 Injection in Patients Undergoing Unilateral Total Knee Arthroplasty
Brief Title: Study to Evaluate Safety/Efficacy of a Single Preop Dose of AYX1 Injection to Treat Pain After Knee Replacement Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adynxx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADYX-004
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Post-surgical Pain
Keywords: post-surgical pain; total knee arthroplasty; total knee replacement
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AYX1 Injection 660 mg/6 mL (Experimental): Single Intrathecal (spinal) administration of AYX1 Injection (660 mg in 6 mL) just prior to intrathecal administration of spinal anesthetic for knee surgery.
  Interventions: Drug: AYX1 Injection 660 mg/6 mL
- Placebo Injection 6 mL (Placebo Comparator): Single Intrathecal (spinal) administration of Placebo Injection (6 mL) just prior to intrathecal administration of spinal anesthetic for knee surgery
  Interventions: Drug: Placebo Injection 6 mL

INTERVENTIONS:
Drug: AYX1 Injection 660 mg/6 mL — 6 mL solution for intrathecal injection with 660 mg of AYX1 (Brivoligide)
  Other Names: Brivoligide 660 mg/6 mL
  Arms: AYX1 Injection 660 mg/6 mL
Drug: Placebo Injection 6 mL — 6 mL solution for intrathecal injection; vehicle formulation designed to mimic AYX1 Injection (with no active drug)
  Arms: Placebo Injection 6 mL

SUMMARY:
The objectives of this study are to evaluate the safety and analgesic efficacy of a single preoperative intrathecal administration of AYX1 Injection in patients undergoing unilateral total knee arthroplasty.

DETAILED DESCRIPTION:
This is a multi-center, Phase 2, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of AYX1 Injection administered intrathecally before surgery in patients undergoing primary unilateral total knee arthroplasty (TKA). Subjects will be randomized on the day of surgery to receive either intrathecal AYX1 Injection or intrathecal placebo just prior to surgery. Study assessments will be conducted during the inpatient period through 48 hours; follow-up visits will be performed through Study Day 90.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo primary unilateral TKA with spinal anesthesia for painful osteoarthritis without congenital knee pathology
* American Society of Anesthesiologists Physical Status Classification System ≤ 3
* Medically stable as determined by the Investigator based on pre-study medical history, physical examination, clinical laboratory tests, and 12-lead electrocardiogram (ECG) findings
* Body Mass Index of 18-45 kg/m2
* Stable medical regimen for at least 1 week before randomization
* Able to read and understand study instructions in English, and willing and able to comply with all study procedures

Exclusion Criteria:

* More than 2 other current focal areas of pain, any pain areas greater in intensity than the target knee, or any other active chronic pain conditions that would compromise operative knee pain evaluation
* Inflammatory arthridities (e.g., rheumatoid arthritis, lupus, ankylosing spondylitis, psoriatic arthritis), with the exception of clinically stable/non-active gout that does not affect the knee and does not interfere with walking
* Surgery in either knee within 3 months prior to randomization, or surgery in either knee greater than 3 months prior to randomization with residual symptoms that would interfere with post-TKA study assessments; use of cryoneurolysis (including Iovera) on the current operative knee region within the 6 months prior to randomization and/or at any time through the duration of the study
* Planned use of general anesthesia or potent inhalational agents, peripheral nerve block (e.g., femoral nerve block), neuroaxial (intrathecal or epidural) opioids, preoperative extended release/long acting opioids, or any use of ketamine preoperatively and/or at any time through the duration of the study
* Use of more than 40 mg per day (on average) of oral morphine or its equivalent within 1 month prior to randomization
* Use of gabapentin or pregabalin within 1 week prior to randomization or planned use post-operatively through Day 28
* Use of systemic corticosteroids (IV or oral) within 3 months prior to randomization through Day 28; planned use of intra-articular steroid injections in the operative knee from the time of randomization through Day 28
* Current neurologic disorder, which could confound the assessment of pain (e.g., Parkinson's, Multiple Sclerosis)
* Untreated or inadequately treated (in the opinion of the Investigator) active depression
* Mini Mental State Exam score < 24 at screening
* History of alcohol-related complications within 1 year of randomization including, but not limited to, alcoholic withdrawal seizures, hallucinations, delirium tremens or detoxification treatment
* Known or suspected history of illicit drug use within 1 year before randomization, or current or planned use of marijuana (including medical approved use) within 1 month before randomization and/or through the duration of the study
* Any confirmed malignancy within the past year, with the exception of basal cell carcinoma or uncomplicated or stable skin cancers documented to not require further or immediate treatment
* Women who are pregnant or nursing
* Previous participation in any study involving AYX1 Injection

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Mean pain with walking during the 15 meter walk test Day 7 to Day 28 | 7-28 days post-surgery
  Mean pain rating on the Numerical Rating Scale (NRS) with walking during the 15 meter walk test during the outpatient period from Day 7 to Day 28

SECONDARY OUTCOMES:
Percentage of subjects with NRS pain score ≥ 4 during the 15 meter walk at Day 90 | at 90 days post-surgery
  Percentage of subjects with the Numerical Rating Scale (NRS) pain score ≥ 4 during the 15 meter walk at Day 90
Mean pain rating (NRS) at rest Day 7 to Day 28 | 7-28 days post-surgery
  Mean pain rating with the Numerical Rating Scale (NRS) at rest Day 7 to Day 28
Total use of postoperative opioid medications (morphine equivalents) post-discharge to Day 90 | post-hospital discharge through 90 days post-surgery
  Total use of postoperative opioid medications (morphine equivalents) post-discharge to Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Donald C Manning, MD, PhD, Study Director — Adynxx, Inc.
Locations (9):
- United States (9):
  - Alabama Orthopedic Center, Birmingham, Alabama
  - Shoals Medical Trials, Sheffield, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - CORE Orthopaedic Medical Center, Encinitas, California
  - Pensacola Research Consultants, Pensacola, Florida
  - Phoenix Clinical Research, Tamarac, Florida
  - Mississippi Sports Medicine, Jackson, Mississippi
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Antria, Inc., Indiana, Pennsylvania

IPD SHARING:
Plan to Share IPD: No